CLINICAL TRIAL: NCT01693991
Title: Randomized Controlled Trial of the Meaning-Making Intervention (MMi) in Patients Newly Diagnosed With Advanced Cancer: A Pilot Study
Brief Title: Randomized Controlled Trial of the Meaning-Making Intervention (MMi)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Melissa Henry, Psychologist, Jewish General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 258431
Record Dates: First submitted 2012-09-18; First posted 2012-09-26 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meaning-Making intervention (MMi) (Experimental): Patients in this arm will be receiving the Meaning-Making intervention (MMi) as per intervention manual (Lee, 2006).
  Interventions: Behavioral: Meaning-Making intervention (MMi)
- Empathic visitor (Placebo Comparator): This person will provide the basic ingredients fostering a good therapeutic relationship (i.e., trust, warmth, empathy, neutrality and authenticity) without further intervention or probing. The empathic visitor will be specifically instructed to avoid initiating discussions about meaning (e.g., how the patient interprets his feelings and thoughts, understands his/her illness and meaning in life), and focus discussions on what is currently happening (rather than on the interface between past and present).
  Interventions: Behavioral: Empathic visitor
- Control Group (No Intervention): Patients in this group will only be receiving treatment as usual.

INTERVENTIONS:
Behavioral: Meaning-Making intervention (MMi) — MMi and attention control sessions will take place weekly for 3 weeks at the patient's home or hospital, as the patient prefers. We will try to limit delays to no more than 1 week if needed (e.g., for recovery from treatment side-effects), but because the feasibility of this schedule is one of the research questions, if more flexibility is required we will not withdraw people from the study if the delay is longer, since a longer intervention period could be incorporated in a full-scale RCT. Dates and duration of each session will be tracked. MMi sessions will be conducted by 2 bilingual mental health professionals (nurse, social worker, or psychologist) with at least 1 year of clinical oncology experience and will be initiated within 1 week after randomization.
  Other Names: MMi
  Arms: Meaning-Making intervention (MMi)
Behavioral: Empathic visitor — This person will provide the basic ingredients fostering a good therapeutic relationship (i.e., trust, warmth, empathy, neutrality and authenticity) without further intervention or probing. The empathic visitor will be specifically instructed to avoid initiating discussions about meaning (e.g., how the patient interprets his feelings and thoughts, understands his/her illness and meaning in life), and focus discussions on what is currently happening (rather than on the interface between past and present).
  Arms: Empathic visitor

SUMMARY:
Research questions: Pilot study research questions: Primary: 1)Can we recruit a sufficient number (i.e., at least 60 patients over 9 months) and retain a sufficient proportion of both men and women (i.e., at least 80% at 2, 4, or 6 months post-randomization) with advanced cancer in all 3 trial arms to allow completion of a full study in 4 years?; 2)Is MMi acceptable: to a general ACP? to both men and women?; Secondary: 1)Is it feasible to complete the intervention in 3-4 weeks? 2)How long is it feasible to test MMi effects: 2, 4 or 6 months post-randomization(retention rate=80%)? 3)Which recruitment strategies are most helpful? 4)What sample size is needed for a full study? Full-study research questions: Primary: Does adding the MMi to usual care (experimental group or EG) enhance meaning in life among newly diagnosed ACP, compared with those receiving usual care plus meetings with an empathic non-professional visitor (i.e., attention-control group or AC) or usual care alone (UC), at x months post-randomization? (time determined in pilot) "Meaning in life" (primary outcome) is defined as the belief that one's life has significance and purpose (i.e., global meaning) and "newly diagnosed ACP" is defined as the 6 months after first occurrence of, progression toward, or recurrence of stage III or IV cancer (TNM classification system). Secondary: In our future full-study, we plan to evaluate MMi effects on secondary outcomes such as existential wellbeing (MQOL existential wellbeing) and posttraumatic growth (Post-Traumatic Growth Inventory). We also plan to test a theoretical model where sense of meaning in life has a protective (moderating) effect on tertiary outcomes such as physical QoL (MQOL physical subscale), anxiety and depression (Hospital Anxiety and Depression Scale (HADS)), and overall QoL (MQOL Total) in EG patients. Methodology: RCT pilot study with 60 newly diagnosed ACP (stages III or IV) within 2 months of referral and 6 months of randomization, assigned randomly to: (1) EG, (2) AC, or (3) UC. Patients will complete self-report questionnaires (including outcome measures, as well as sociodemographic and medical variables) at 2, 4 and 6 months post-randomization.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria: 1) Diagnosed with advanced cancer (stage III or IV --TNM classification system; 117); first occurrence, progression or recurrence) of any type of solid tumour <2 months at referral and <6 months at randomization. 2) Willing to participate in weekly MMi or AC sessions. 3) >18 years. 4) Alert and capable of giving free and informed consent. 5) Able to speak and read English or French. Exclusion Criteria: 1) Karnofsky Performance Status (KPS) score <60 (rated by referring oncologists/nurses or Research Coordinator (RC)) or expected survival <6 months according to clinical judgment. 2) Currently receiving radiotherapy (Rx) treatment (although these patients can be reassessed after Rx). Patients will only be included in the study when they have recovered from severe side-effects from Rx and when they feel they can participate in the study. Severe side-effects are defined as a score of 3 or 4 on any of the site-specific toxicity markers of the Eastern Cooperative Oncology Group (ECOG) Common Toxicity Criteria or with more than 3 markers with a score of 2 (moderate side-effects), as evaluated by the treating physician (in consultation with the radiotherapist. 3) Suicidal. Present a score of ≥2 on the Beck Depression Inventory (BDI) suicide item (item #9), administered by the RC or RA during the consent meeting. 4) Known diagnosis of schizophrenia or schizoaffective disorder. 5) Planning a trip within 2 months that would interrupt delivery of the MMi or AC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 months post randomization
  1. Can we recruit a sufficient number (i.e., 60 patients over 9 months or 6.7 per month) of newly diagnosed advanced cancer patients? AND
  2. Can we retain a sufficient proportion of both men and women (i.e., at least 80%) with advanced cancer in all 3 trial arms to allow completion of a full study in 4 years?
Acceptability | 2 months post-randomization
  Is the MMi acceptable to at least 80% of men and women with advanced cancer, as indicated by 80% positive responses on the Pilot-Study Questionnaire (PSQ; adapted from the CSQ-8; Attkisson & Zwick, 1982) Q#7 (score 3 or 4), Q#8, and Q#9 (score 5, 6 or 7).
  PSQ Q#7: Would you recommend those types of meetings to other people in your situation? 1= no, definitively not; 2= no, I don't think so; 3= yes, I think so; 4= yes, definitively PSQ Q#8: Were the meetings acceptable? PSQ Q#9: On the whole, how positive or negative was your experience of the meetings? 1= Totally negative; 2= Very negative; 3= A little negative; 4= Neutral; 5= A little positive; 6= Very positive; 7= Totally positive

SECONDARY OUTCOMES:
Timing of the intervention | 2 month post-randomization
  Will at least 95% of EG and AC patients complete the intervention in 3-4 weeks?
Primary evaluation time | 6 months post-randomization
  Which evaluation time should be primary, 2, 4 or 6 months post-randomization, based on an acceptable retention rate of 80%?
Recruitment strategies | 2 months post-randomization
  Which recruitment strategies are most effective, defined as the strategies recruiting the largest % of participants. Strategies recruiting <5% of participants will be considered unhelpful. All participants will be queried as to how they found out about the study. Recruitment strategies will include: being recruiting directly through the treating team, posted ads in recruiting oncology clinics, use of local media (newspaper and radio interviews), and creation of a website linked with the Jewish General Hospital and the McGill University Health Centre.
Sample size calculation for the full study | 2 months post-randomization
  What is the 80% upper confidence interval for the standard deviation at baseline?

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Henry, Ph.D., Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital; and McGill University; S Robin Cohen, Ph.D., Principal Investigator — Lady Davis Institute for Medical Research, Jewish General Hospital; and McGill University
Locations (2):
- Canada (2):
  - McGill University Health Centre, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec